CLINICAL TRIAL: NCT05841251
Title: Phenylephrine Versus Tranexamic Acid to Control Bleeding in Patients Undergoing Inferior Turbinoplasty by Coblation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Aboulfotouh Mohammed, lecturer of Anesthesia and icu, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 27111344
Record Dates: First submitted 2023-04-11; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Intraoperative Bleeding; Coblation Turbinoplasty
MeSH Terms: conditions — Blood Loss, Surgical

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- phenylephrine (Active Comparator): phenylephrine-soaked pack will be applied after induction of surgery and intubation.
  Interventions: Drug: Topical Phenylephrine Solution
- tranexamic acid (Active Comparator): Single intravenous dose of tranexamic acid 15 mg/kg will be given in 100 mL normal saline over 10 minutes.
  Interventions: Drug: intravenous tranexamic acid

INTERVENTIONS:
Drug: Topical Phenylephrine Solution — phenylephrine-soaked pack using the whole 5 ml of the solution provided with.5% phenylephrine will be applied after induction of surgery and intubation, 15 minutes before surgery. 100 ml of normal saline will be given.
  Arms: phenylephrine
Drug: intravenous tranexamic acid — patients will receive intravenous Single dose of tranexamic acid 15 mg/kg in 100 mL normal saline over 10 minutes. Saline-soaked pack will be applied.
  Arms: tranexamic acid

SUMMARY:
Coblation is a unique method of delivering radio frequency energy to the soft tissue for applications in otolaryngology. It induces reduction of the inferior turbinate by vaporizing and destroying the soft erectile tissue. The volume reduction and tissue fibrosis are immediate and sustainable. Bleeding from the vascular capillary beds of the sinonasal mucosa compromises the surgical field and increases operative time and risk of complications. In this study we try to assist hemostasis with a multifaceted approach, including use of topical vasoconstrictors "phenylephrine" and systemic antifibrinolytic agent "tranexamic acid".

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I and II
* Scheduled patients for Coblation Turbinoplasty surgery with inferior turbinate hypertrophy

Exclusion Criteria:

* Known allergy to study drugs.
* History of coagulopathy or bleeding disorders.
* Patients with hypertension or ischemic heart disease.
* patients on anticoagulants, antiplatelets or NSAIDs
* history of deep vein thrombosis, stroke or peripheral vascular disease.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
surgical field scale | intraoperativel
  the intraoperative surgical site bleeding using the surgical field scale as follows: 0 = No bleeding
  1. = Minimal bleeding: Not a surgical nuisance and no suction required
  2. = Mild bleeding: Occasional suction required, but does not affect dissection
  3. = Moderate bleeding: Slightly compromises surgical field, frequent suction required
  4. = Severe bleeding: Significantly compromises surgical field, frequent suction required, bleeding threat field just after removal of suction
  5. = Massive bleeding: Prevent dissection.

SECONDARY OUTCOMES:
Volume of Blood loss | intraoperative
Duration of surgery | the duration from induction of anesthesia till extubation
Avoidance of postoperative nasal packing | immediately after the surgey
  if the patient can be spared from postoperatiove nasal pack inserted for controllling bleeding
Intra-operative and Postoperative complications | intraoperative and 24 hours postoperative
  Complications such as nausea, vomiting, hypotnsion, hypertension, hemorraghic or thrombotic manifestations for 24 hours